CLINICAL TRIAL: NCT04947410
Title: Intestinal Dysbiosis During Obstructive Sleep Apnea Syndrome : Impact of Continuous Positive Airway Pressure (CPAP) - A Randomized Controlled Trial Versus Nasal Dilators
Brief Title: Intestinal Dysbiosis During Obstructive Sleep Apnea Syndrome
Acronym: DYNAMIC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulty
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 38RC19.057
Record Dates: First submitted 2021-06-23; First posted 2021-07-01 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Obstructive Sleep Apnea Syndrome; Gut Microbiota
Keywords: intermittent hypoxia; intestinal dysbiosis
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: 2 interventional groups (15 OSAS patients into "CPAP group" versus 15 OSAS patients into "nasal dilators group") are evaluated in parallel against a control group (15 Non-OSAS Patients)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OSAS Patients treated with CPAP (Active Comparator): Patients with OSAS will have 1 in 2 chance of being randomized into "CPAP group"
  Interventions: Device: CPAP or nasal dilators
- OSAS Patients treated with nasal dilators (Sham Comparator): Patients with OSAS will have 1 in 2 chance of being randomized into "nasal dilators group"
  Interventions: Device: CPAP or nasal dilators
- Non OSAS Patients (No Intervention): Non OSAS Patients will be the parallel control group

INTERVENTIONS:
Device: CPAP or nasal dilators — CPAP = active comparator nasal dilators = placebo comparator
  Arms: OSAS Patients treated with CPAP; OSAS Patients treated with nasal dilators

SUMMARY:
Obstructive Sleep Apnea Syndrome (OSA) is one of the most common chronic diseases and is associated with prognostic cardiovascular and metabolic co-morbidities. OSAS is the recurrence of complete (apnea) or partial (hypopnea) collapse of the upper airway during sleep resulting in sleep fragmentation and chronic intermittent hypoxia (ICH) which are the major determinants of cardiovascular and metabolic complications including type 2 diabetes, obesity and non-alcoholic fatty liver. These comorbidities are associated with a change in intestinal microbial ecology. In most cases, there is a reduction in bacterial genetic diversity and more or less specific signatures of cardiovascular and metabolic diseases, making it possible to envisage personalized and innovative therapeutic treatments. In animals exposed to intermittent hypoxia, there is local hypoxia that increases intestinal permeability, produces a reduction in microbiota diversity and favors microbial species that are at the origin of pro-inflammatory factors. Continuous Positive Airway Pressure (CPAP) is the standard treatment for OSA. Its effect on the intestinal microbiota has not yet been evaluated.

DETAILED DESCRIPTION:
Background :

Obstructive Sleep Apnea Syndrome (OSAS) is one of the most common chronic diseases associated with cardiovascular and metabolic comorbidities (high blood pressure, type 2 diabetes, obesity and non-alcoholic fatty liver disease) that make it a prognosis.

These comorbidities are associated with a change in intestinal microbial ecology. In most cases, there is a reduction in bacterial genetic diversity and more or less specific signatures of cardiovascular and metabolic diseases which make it possible to envisage personalized and innovative therapeutic treatments.

In animals exposed to intermittent hypoxia, there is a local hypoxia that increases intestinal permeability, produces a reduction in microbial diversity, and favors microbial species that cause the secretion of pro-inflammatory factors.

Continuous Positive Airway Pressure (CPAP) is the gold standard for OSAS treatment. Its effect on the gut microbiota has never been evaluated.

The data will be totally original in the field. The impact of this study can be major in allowing to propose pre/probiotics or drug treatments modulating intestinal dysbiosis during OSAS, combined or not with CPAP.

Objective:

The principal objective of the study is to compare gut microbiota changes (diversity and composition : relative abundance of different phyla, genera, families, alpha and beta diversity...) after 3 months of effective CPAP versus 3 months of placebo (nasal dilators), in patients with Obstructive Sleep Apnea Syndrome.

The second objectives

Methods :

OSAS patients (with AHI > 30 / hour) will be screened in EFCR Service, Pneumology Department or Sleep Laboratory and proposed the study. If eligible they will be then followed over 3 months with 2 visits (inclusion visit at J0 and follow-up visit at 3 months). After the inclusion visit (J0) OSAS patients will be randomized for their treatment into "CPAP group" (effective CPAP treatment) or "nasal dilators group" (placebo treatment) for 3 months.

The same assessments will be carried out at J0 and 3 months.

Healthy volunteers (with no OSAS) will be the control group. They will be recruited by ad. They will carry out the assessments of inclusion visit (J0) only and compared then to the group of OSAS patients.

ELIGIBILITY:
Inclusion Criteria:

Non-SAOS Group :

* Men or women aged 18 to 70
* Subject without any OSAS
* Subject with Body Mass Index < 30 kg/m2
* Subject who has given their free and informed consent in writing
* Subject affiliated to the French social security system (or equivalent)

SAOS Group :

* Men or women aged 18 to 70
* Subject with OSAS (Apnea-hypopnea index > 30/hour)
* Patient with CPAP indication and untreated at baseline
* Subject with Body Mass Index < 30 kg/m2
* Effective contraception for women of childbearing age (progestational or estrogen-progestin hormonal contraceptives (pill, ring, transdermal patch), intrauterine devices or definitive sterilization)
* Subject who has given their free and informed consent in writing
* Subject affiliated to the French social security system (or equivalent)

Exclusion Criteria:

* Patient with resistant hypertension (PA ≥ 140/90 mmHg despite taking at least 3 drugs of different therapeutic classes at near maximal dose, including a diuretic)
* Infection, progressive neoplasia, unstable cardiovascular pathologies, metabolic or intestinal pathologies
* Taking of pre/probiotics and/or antibiotics in the 6 months prior to inclusion
* Major sleepiness in at-risk populations for whom the introduction of treatment by CPAP equipment is mandatory and rapid (truck drivers, crane operators ...) according to the investigator
* Patient with major desaturations during its polysomnographic diagnostic recording (≥ 2h with O2 saturation <90% on total sleep time)
* Patient with high daytime sleepiness (Epworth score > 15)
* Contraindication to the implementation of a CPAP treatment for the SAOS group
* Contraindication to perform a subcutaneous biopsy (subject with hypersensitivity to a known local anaesthetic, abdominal skin lesion ...)
* Drastic diet (vegetarian, vegan, pescetarian), food allergies
* Subject referred to in Articles L1121-5 to L1121-8 of the CSP (pregnant woman, parturient, mother who is breast-feeding, person deprived of liberty by judicial or administrative decision, legally protected person)
* Subject being in an exclusion period of another study or ongoing participation in a drug study
* Patient likely, in the opinion of the investigator, not to be cooperative or respectful of the obligations inherent to participation in the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-11-23 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Diversity and composition of the microbiota (relative abundance of different phyla, genera, families, alpha (intra-sample) and beta (inter-sample) diversity ...) | 3 months
  This analysis will compare changes in intestinal microbiota after 3 months of effective CPAP versus 3 months of placebo CPAP (sham-CPAP )

SECONDARY OUTCOMES:
Comparison of the intestinal microbiota between non-OSAS subjects and OSAS patients (before treatment with CPAP or nasal dilators) | At inclusion visit (V1)
  Comparison of the diversity and composition of the microbiota (relative abundance of different phyla, genera, families, etc.) between the two groups (OSAS and non-OSAS).
Correlation between changes in arterial blood pressure and microbiota changes between OSAS and non-OSAS, and then between CPAP and nasal dilators, after 3 months of treatment only for OSAS patients | 3 months
  Correlation between mean, systolic and diastolic 24 hours (day and night) arterial pressures, measured by 24-hours ambulatory recording, and modifications of the microbiota by OSAS and then by CPAP or nasal dilators
Correlation between changes in lipid and carbohydrate profiles and changes in microbiota between OSAS patients and non-OSAS subjects, then between CPAP and nasal dilators groups after 3 months of treatment | 3 months
  Correlation between changes in fasting blood glucose, glycated hemoglobin (HbA1c), total cholesterol, HDL-Cholesterol, LDL-Cholesterol, triglycerides and modifications of the microbiota by OSAS and then by CPAP or nasal dilators
Comparison of markers of inflammation, senescence and remodeling of adipose tissue between OSAS and non-OSAS, and then between CPAP and nasal dilators after 3 months of treatment | 3 months
  Senescence markers, adipose RNA, cytokines, immunophenotyping of macrophages

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, PhD, Principal Investigator — University Grenoble Hospital